CLINICAL TRIAL: NCT06998550
Title: Patient Experiences and the Role of Team Structures in Pulmonary Rehabilitation in Türkiye: The PRETTY Study - A National, Multicenter, Cross-Sectional Observational Study
Brief Title: Patient Experiences and the Role of Team Structures in Pulmonary Rehabilitation in Türkiye
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, PhD, Saglik Bilimleri Universitesi
Other Study IDs: PRETTY Study
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease; Pulmonary Rehabilitation
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PatiePatient Group: Individuals Who Completed a Pulmonary Rehabilitation Programnts: Adult patients with a respiratory disease who have completed a pulmonary rehabilitation (PR) program, regardless of the setting (inpatient, outpatient, or home-based).
  Interventions: Other: Patient Satisfaction Questionnaire
- Institutional Representative Group: Pulmonary Rehabilitation Program Coordinators: Healthcare professionals (e.g., physiotherapists, pulmonologists, or allied health staff) who are designated as coordinators or key team members responsible for organizing and managing the pulmonary rehabilitation program in their institution.
  Interventions: Other: Institutional Survey on PR Program Structure and Team Composition

INTERVENTIONS:
Other: Patient Satisfaction Questionnaire — An online survey designed to assess patient experiences and satisfaction levels with pulmonary rehabilitation (PR) programs. The questionnaire covers aspects such as accessibility, communication, program structure, perceived outcomes, and overall satisfaction. It is administered via Google Forms and completed voluntarily by patients who have completed a PR program.
  Groups: PatiePatient Group: Individuals Who Completed a Pulmonary Rehabilitation Programnts
Other: Institutional Survey on PR Program Structure and Team Composition — A structured online questionnaire completed by the designated PR program coordinator or team member. It includes questions on organizational features of the PR program, such as team composition, session frequency, assessment tools, referral and admission
  Groups: Institutional Representative Group: Pulmonary Rehabilitation Program Coordinators

SUMMARY:
The PRETTY Study aims to evaluate patient satisfaction with pulmonary rehabilitation (PR) services across Türkiye and to investigate how satisfaction levels are related to the organizational structures and team compositions of the PR programs. This national, multicenter, cross-sectional observational study will also identify structural and organizational factors that may enhance patient-centered care and promote the standardization of PR services.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age ≥18 years
* Diagnosed with a respiratory condition (e.g., COPD, interstitial lung disease, asthma, bronchiectasis, etc.)
* Completed a structured PR program (minimum duration and frequency as defined by national guidelines or center-specific protocols)
* Willing and able to complete the online Patient Satisfaction Questionnaire
* Able to provide informed consent

Patient Exclusion Criteria:

* Ongoing participation in a PR program (only completed cases will be included)
* Inability to complete the questionnaire due to cognitive or language barriers without a caregiver

Coordinator Inclusion Criteria:

* Officially designated as the PR program coordinator or responsible team member
* Affiliated with a healthcare institution (public, university-affiliated, or private) in Türkiye that provides PR services
* Willing to complete the Institutional Survey Form regarding team structure, service delivery, and organizational characteristics
* Authorized by the institution to provide structural data related to the PR unit

Coordinator Exclusion Criteria:

* PR services provided on an informal or ad-hoc basis without a designated team or structure
* Institutions not offering a structured PR program

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group/Cohort 1 (Label): Patient Group Description: Adults with respiratory disease who have completed a PR program and will complete the Patient Satisfaction Questionnaire.
  Group/Cohort 2 (Label): Program Coordinator Group Description: Healthcare professionals responsible for PR program coordination who will complete the Institutional Survey Form about organizational and team structures.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Questionnaire | Within 4 weeks after completion of the pulmonary rehabilitation program
  An online survey designed to assess patient experiences and satisfaction levels with pulmonary rehabilitation (PR) programs. The questionnaire covers aspects such as accessibility, communication, program structure, perceived outcomes, and overall satisfaction. It is administered via Google Forms and completed voluntarily by patients who have completed a PR program.
Institutional Survey on PR Program Structure and Team Composition | Within 4 weeks after completion of the pulmonary rehabilitation program
  A structured online questionnaire completed by the designated PR program coordinator or team member. It includes questions on organizational features of the PR program, such as team composition, session frequency, assessment tools, referral and admission criteria, and program setting (inpatient, outpatient, or home-based). This survey aims to document the structural diversity of PR services across different healthcare institutions.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided